CLINICAL TRIAL: NCT05845619
Title: Implementing a Risk Score to Facilitate Enhanced Adherence Support for Pregnant and Postpartum Women at Risk of Viremia
Brief Title: Enhanced Virologic Monitoring for Pregnant and Postpartum Women With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K01MH119910 (NIH); K01MH119910 (NIH)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; Viremia; Pregnancy Related
MeSH Terms: conditions — HIV Infections; Viremia

STUDY DESIGN:
Intervention Model Description: Pilot study participants will be compared to historical controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilot (Experimental)
  Interventions: Behavioral: Enhanced virologic monitoring
- Controls - prospectively enrolled (No Intervention)
- Controls - abstracted from records (No Intervention)

INTERVENTIONS:
Behavioral: Enhanced virologic monitoring — The pilot intervention will include the following components:
  1. More frequent viral load collection: Participants who enroll in the first 3 months of the pilot study period will be eligible for a 3-month follow-up visit and will have viral load assessed again at that time.
  2. Rapid return of viral load results: Mentor mothers (peer counselors) will be trained to return viral load results to patients. Viral loads will will be processed with GeneXpert point of care technology.
  3. Enhanced viral load counseling: Mentor mothers will reinforce adherence with all patients with undetectable levels via scripted messaging to reward and encourage healthy behavior. For those with any detectable levels, mentor mothers will be trained to provide targeted counseling with scripted messaging according to viral load level (undetectable, low-level viremia (50-1000), high viral load (>1000)).
  Arms: Pilot

SUMMARY:
The goal of this study is to learn about supporting pregnant and postpartum women living with HIV with treatment adherence. The investigators will conduct a pilot study of an intervention that includes peer counseling about viral load levels and rapid delivery of viral load results. The investigators will evaluate the feasibility of the intervention, and will assess whether it improves viral suppression 6 months following the intervention, compared to historical controls.

DETAILED DESCRIPTION:
The investigators will examine the use of more frequent virologic monitoring with enhanced communication around low-level viremia as a strategy to identify and support pregnant and postpartum women at risk of virologic failure. Virologic monitoring itself can reinforce adherence in stable patients, and more frequent monitoring can detect potential adherence challenges early. Notably, low-level viremia is a strong predictor of subsequent virologic failure, and the lowest level associated with perinatal transmission is not known.

The pilot study will run for 6 months at 4 Ministry of Health facilities in Kisumu County, Kenya; 275 participants will be enrolled. Prior to the pilot study, 125 controls will be enrolled prospectively, and 150 controls will be abstracted from records from the prior year.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV
* On antiretroviral treatment
* Either pregnant in the 3rd trimester, OR, postpartum within 6 months of delivery

Exclusion Criteria:

* n/a

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Murnane, PhD, Principal Investigator — University of California, San Francisco
Locations (4):
- Kenya (4):
  - Lumumba Sub County Hospital, Kisumu
  - Nyakach County Hospital, Nyakach
  - Ahero County Hospital, Nyando
  - Rabuor Sub county Hospital, Nyando

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murnane PM, Ouma S, Onyango R, Mukand N, Thapar I, Odhiambo F, Kabami J, Bukusi EA, Cohen CR, Ayieko J. Engaging Mentor Mothers in Rapid Return of Viral Load Results to Pregnant and Postpartum Women Living with HIV: An Implementation Pilot Study. AIDS Behav. 2025 Dec 23. doi: 10.1007/s10461-025-04987-2. Online ahead of print. PMID 41432869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 550 participants
Pre-assignment Details: There was no pre-assignment procedure
Groups:
- Controls - Prospectively Enrolled; Controls - Abstracted From Records: routine care
Period: Overall Study
Arm/Group | Pilot | Controls - Prospectively Enrolled | Controls - Abstracted From Records
Started | 275 | 125 | 150
Completed | 273 | 123 | 149
Not Completed | 2 | 2 | 1
Not completed — duplicate enrollment | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot | Controls - Prospectively Enrolled | Controls - Abstracted From Records | Total
Number analyzed (Participants) | 273 | 123 | 149 | 545
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 34] | 30 [27 to 34] | 31 [27 to 36] | 30 [26 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 123 | 149 | 545
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 273 | 123 | 149 | 545
Region of Enrollment [Number; unit: participants]
  Kenya | 273 | 123 | 149 | 545
Viral load in prior 12 months [Count of Participants; unit: Participants] — Values were collected from records only, no study participant interaction. (Suppression=good; non-suppression=not good; missing=unknown)
  Participants
    Suppressed viral load (per clinical records) | 175 | 82 | 94 | 351
    Not suppressed viral load (per clinical records) | 47 | 21 | 18 | 86
    No record (missing) | 51 | 20 | 37 | 108

OUTCOME MEASURES:

1. Primary Outcome: Plasma HIV RNA >50 Copies/mL
Description: Plasma HIV RNA >50 copies/mL. Data will be collected from clinical records only, no participant interaction. If >1 viral load is collected during the time frame below, the first will be used.
Time Frame: Within 6 months after study engagement (i.e., after pilot study participation; after the enrollment visit for prospectively enrolled controls; after the date of eligibility for controls from records)
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Pilot: Enhanced virologic monitoring
Arm/Group | Pilot | Controls - Prospectively Enrolled | Controls - Abstracted From Records
Number analyzed (Participants) | 273 | 123 | 149
Participants | 34 | 13 | 15
Statistical Analysis 1: Comparison: Pilot vs Controls - Prospectively Enrolled; In this pilot study, we hypothesized that pilot participants would have a reduced risk of viremia 6 months after the intervention compared to controls; Test type: Superiority — There was no power calculation because this was a pilot study; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.83 to 1.76] — Numerator: pilot; denominator: prospective controls
Statistical Analysis 2: Comparison: Pilot vs Controls - Abstracted From Records; Test type: Superiority — No power calculation, pilot study; p = 0.41, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.73 to 2.14]

ADVERSE EVENTS:
Time Frame: Prospectively enrolled controls had only one cross sectional visit. Among 273 pilot participants, 124 had only a baseline cross sectional visit and 149 had both a baseline visit and a 3 month follow up visit. (this was a 6-month pilot implementation study at the facilities, and thus only those enrolled during the first 3 months reached the period in which a 3 month follow- up was possible)
Description: We followed the clinicaltrials.gov definition of an adverse event.
Arm/Group | Pilot | Controls - Prospectively Enrolled | Controls - Abstracted From Records
All-Cause Mortality (participants affected / at risk) | 0/273 | 0/123 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/273 | 0/123 | 0/149
Other Adverse Events (participants affected / at risk) | 0/273 | 0/123 | 0/149

LIMITATIONS AND CAVEATS:
This was a pilot study, and therefore not powered to detect statistically significant differences between intervention and control. Additionally, participants were not randomized and may have different baseline risks for subsequent viremia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT05845619/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT05845619/ICF_000.pdf